CLINICAL TRIAL: NCT01932437
Title: A Randomized, Double-Blind, Single Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of Single Intramuscular Doses of ETI-204 in Adult Volunteers
Brief Title: Intramuscular Dose-Escalation Study With ETI-204 in Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elusys Therapeutics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: AH106
Record Dates: First submitted 2013-08-02; First posted 2013-08-30 (Estimated); Results first posted 2019-05-01 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-04

CONDITIONS: Inhalational Anthrax
Keywords: Monoclonal antibody, ETI-204, IM, safety, PK, immunogenicity
MeSH Terms: conditions — Inhalation anthrax | interventions — obiltoxaximab

STUDY DESIGN:
Intervention Model Description: Dose escalation study
Who Masked: Participant, Care Provider, Investigator
Masking Description: The investigator, clinical research unit staff, and subjects will be blinded to treatment assignment. The randomization list will be made available to the pharmacist preparing study drug.
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): 3 subjects will receive an IM dose of 4 mg/kg ETI-204, administered as two injections with a maximum volume of 2 mL at each injection site.
  1 subject will receive an IM dose of ETI-204-placebo in an identical fashion.
  Interventions: Biological: ETI-204; Other: Placebo
- Cohort 2 (Experimental): 6 subjects will receive an IM dose of 8 mg/kg ETI-204, administered as two injections with a maximum volume of 4 mL at each injection site.
  2 subjects will receive an IM dose of ETI-204-placebo in an identical fashion.
  Interventions: Biological: ETI-204; Other: Placebo
- Cohort 3 (Experimental): 6 subjects will receive an IM dose of 16 mg/kg ETI-204, administered at four sites, with administration of 4 mL at one site and the remaining volume given in three additional injections with a maximum volume of 4 mL at each injection site.
  2 subjects will receive an IM dose of ETI-204-placebo in an identical fashion.
  Interventions: Biological: ETI-204; Other: Placebo
- Cohort 4 (Experimental): 6 subjects will receive an IM dose of 20 mg/kg ETI-204, administered at up to five sites, with the injection volume distributed equally between injections and a maximum volume of 4 mL per injection site.
  2 subjects will receive an IM dose of ETI-204-placebo in an identical fashion.
  Interventions: Biological: ETI-204; Other: Placebo
- Cohort 5 (Experimental): 6 subjects will receive an IM dose of 24 mg/kg ETI-204, administered at up to six sites, with administration of 5 mL at one site and the remaining volume given in up to five additional injections distributed equally with a maximum volume of 4 mL per injection site.
  2 subjects will receive an IM dose of ETI-204-placebo in an identical fashion.
  Interventions: Biological: ETI-204; Other: Placebo

INTERVENTIONS:
Biological: ETI-204 — monoclonal antibody
  Other Names: Obiltoxaximab
Other: Placebo — Placebo for ETI-204

SUMMARY:
This study is to evaluate the safety, local tolerability, pharmacokinetics (PK) and immunogenicity of escalating single intramuscular (IM) doses of ETI-204 in healthy volunteers

DETAILED DESCRIPTION:
Following completion of a Screening visit subjects will arrive at the clinic on Day -1. On Day 1, subjects will be randomized in a 3:1 ratio to receive an IM dose of either ETI-204 or matching placebo, respectively:

Cohort 1: 4 subjects randomized to 4 mg/kg ETI-204 or matching placebo Cohort 2: 8 subjects randomized to 8 mg/kg ETI-204 or matching placebo Cohort 3: 8 subjects randomized to 16 mg/kg ETI-204 or matching placebo Cohort 4: 8 subjects randomized to 20 mg/kg ETI-204 or matching placebo Cohort 5: 8 subjects randomized to 24 mg/kg ETI-204 or matching placebo

Study drug will be injected bilaterally into the vastus lateralis muscles, with the subject in a supine position. A separate syringe with a 21-gauge,1.5-inch needle will be used for each injection. The number of injections and injection volume will increase with increasing dose allowing for an assessment of increasing IM ETI-204 doses and the tolerability of a larger number of injections and larger injection volume.

Subjects will be pretreated with 50 mg oral diphenhydramine approximately 30 minutes prior to administration of study drug.

Subjects will be discharged from the study facility on Day 4 following completion of study assessments and will return to the study facility for additional visits on Days 7, 10, 15 (±3 days), 29 (±3 days), 43 (±3 days), and 71 (±4 days).

Decisions to dose-escalate will be made by the investigator(s) in conjunction with the sponsor and will be based solely on the available safety and local tolerability data up to and including Day 4.

ELIGIBILITY:
Inclusion Criteria:

1. Females or males ≥18 years of age;
2. All females regardless of childbearing potential must have a negative serum beta human chorionic gonadotropin (β-hCG) pregnancy test at Screening and Day -1;
3. Females of childbearing potential (i.e., not postmenopausal or surgically sterile) must agree to practice abstinence or to use a medically accepted method of contraception from the time of Screening through 30 days after the final study visit. Acceptable methods of contraception include diaphragm/cervical cap with spermicide; sponge with spermicide; condom with spermicide; or intrauterine device with condom or spermicide. The following contraceptive methods are acceptable only when used with a condom and spermicide: birth control pills, birth control patches, vaginal ring, hormone under the skin, or hormone injections;
4. Postmenopausal females, defined as females who have had amenorrhea for at least 12 months either naturally or following cessation of all exogenous hormonal treatments, and have a follicle stimulating hormone level of >40 mIU/mL at Screening;
5. Females who have undergone surgical sterilization, including hysterectomy, bilateral oophorectomy, bilateral salpingectomy, tubal ligation, or tubal essure;
6. Males must agree to practice abstinence or use a condom with spermicide and to refrain from sperm donation from Screening during the study and for 30 days after the final study visit;
7. Provide written informed consent;
8. Willing to comply with study restrictions.

Exclusion Criteria:

1. Body weight >100 kg;
2. Body mass index ≥32 kg/m2;
3. Pregnant or lactating female;
4. Clinically significant comorbidity that would interfere with completion of the study procedures or objectives, or compromise the subject's safety;
5. Supine systolic blood pressure (BP) ≥150 mmHg or ≤90 mmHg or diastolic BP ≥95 mmHg;
6. Use of H1 receptor antagonists (i.e., antihistamines) within 5 days prior to Day 1;
7. Evidence of drug or alcohol abuse within 6 months of Day 1 as determined by the Investigator;
8. Positive test result for drugs of abuse (with the exception of medically prescribed drugs) at Screening or on Day -1;
9. Positive test for alcohol at Screening, subject to Investigator's discretion. Subjects who test positive for alcohol at Day -1 are excluded from the study;
10. Treatment with an investigational agent within 30 days or 5 half-lives of the investigational agent at Day 1 (whichever is longer);
11. Congenital or acquired immunodeficiency syndrome;
12. Prior solid organ or bone marrow transplant;
13. Positive test for Hepatitis B (surface antigen), Hepatitis C, or human immunodeficiency virus (HIV) at Screening;
14. History of prior treatment for anthrax exposure or prior anthrax infection;
15. Prior immunization with any approved or investigational anthrax vaccine or prior treatment with an investigational anthrax treatment (e.g., ETI-204, raxibacumab, or anthrax immune globulin);
16. Military personnel deployed in 1990 or after, unless the subject can provide documentation demonstrating he or she has not previously received any approved or investigational anthrax vaccine;
17. Use of systemic steroids, immunosuppressive agents, anticoagulants, or anti-arrhythmics within 1 year prior to Day 1. A single short course (i.e., less than 14 days) of systemic steroid therapy is allowed, provided it concluded more than 6 months prior to Day 1;
18. Donation or loss of >500 mL of blood within 30 days or plasma within 7 days of Day 1;
19. Prior stroke, epilepsy, relapsing or degenerative central nervous system disease, or relapsing or degenerative ocular disease;
20. Myocardial infarction or acute coronary syndrome in the past 5 years, active angina pectoris, or heart failure (New York Heart Association scale >1);
21. History of chronic liver disease;
22. Calculated creatinine clearance of <30 mL/min using the Cockcroft-Gault equation;
23. Any clinically significant abnormality, in the Investigator's opinion, on electrocardiogram (ECG) or clinical laboratory tests (hematology, clinical chemistry, or urinalysis) at Screening. Out of range tests may be repeated to confirm;
24. History of allergic or hypersensitivity reaction or hives to other therapeutic antibodies or immunoglobulins;
25. History of any malignant neoplasm within the last 5 years, with the exception of adequately treated localized or in situ non-melanoma carcinoma of the skin (e.g., basal cell carcinoma) or the cervix;
26. Subjects who, in the opinion of the Investigator, are not suitable candidates for enrollment or who may not comply with the requirements of the study.
27. Platelet count <140 K/µL;
28. Prothrombin time/international normalized ratio or activated partial thromboplastin time >1.2 X the upper limit of normal at Screening or Day -1;
29. Poor muscle mass as determined by the Investigator;
30. Family or personal history of a bleeding disorder;
31. History of unexplained bleeding;
32. Use of any anticoagulant or anti-platelet drug for 3 months prior to Screening. At the discretion of the Investigator, daily aspirin may be taken for general health reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-07-26 (Actual); Primary Completion 2014-07-03 (Actual); Study Completion 2014-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex King, MD, Principal Investigator — Covance Clinical Research Unit
Locations (1):
- Covance Clinical Research Unit Inc., Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study started July 26, 2013. Study completed July 03, 2014. Conducted at a Phase 1 Clinical Research Unit
Groups:
- Placebo: Participants received a single intravenous dose of placebo on day 1 followed by a 71 day follow-up.
- ETI-204 4 mg/kg: Participants received a single intravenous dose of ETI-204 4 mg/kg on day 1with a 71-day follow-up period.
- ETI-204 8 mg/kg: Participants received a single intravenous dose of ETI-204 8 mg/kg on day 1 with a 71 day follow-up period.
- ETI-204 16 mg/kg: Participant received a single intravenous dose of ETI-204 16 mg/kg on day 1 with a 71 day follow-up period.
- ETI-204 20 mg/kg: Participants received a single intravenous dose of ETI-204 20 mg/kg on day 1 with a 71 day follow-up period.
- ETI-204 24 mg/kg: Participants received a single intravenous dose of ETI-204 24 mg/kg on day 1 with a 71 day follow-up period.
Period: Cohort 1 - ETI-204 4 mg/kg or Placebo
Arm/Group | Placebo | ETI-204 4 mg/kg | ETI-204 8 mg/kg | ETI-204 16 mg/kg | ETI-204 20 mg/kg | ETI-204 24 mg/kg
Started | 1 | 3 | 0 | 0 | 0 | 0
Completed | 1 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 2 - ETI-204 8 mg/kg or Placebo
Arm/Group | Placebo | ETI-204 4 mg/kg | ETI-204 8 mg/kg | ETI-204 16 mg/kg | ETI-204 20 mg/kg | ETI-204 24 mg/kg
Started | 2 | 0 | 6 | 0 | 0 | 0
Completed | 2 | 0 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 3 - ETI-204 16 mg/kg or Placebo
Arm/Group | Placebo | ETI-204 4 mg/kg | ETI-204 8 mg/kg | ETI-204 16 mg/kg | ETI-204 20 mg/kg | ETI-204 24 mg/kg
Started | 2 | 0 | 0 | 6 | 0 | 0
Completed | 2 | 0 | 0 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 4 - ETI-204 20 mg/kg or Placebo
Arm/Group | Placebo | ETI-204 4 mg/kg | ETI-204 8 mg/kg | ETI-204 16 mg/kg | ETI-204 20 mg/kg | ETI-204 24 mg/kg
Started | 2 | 0 | 0 | 0 | 6 | 0
Completed | 2 | 0 | 0 | 0 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 5 - ETI-204 24 mg/kg or Placebo
Arm/Group | Placebo | ETI-204 4 mg/kg | ETI-204 8 mg/kg | ETI-204 16 mg/kg | ETI-204 20 mg/kg | ETI-204 24 mg/kg
Started | 2 | 0 | 0 | 0 | 0 | 6
Completed | 2 | 0 | 0 | 0 | 0 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: IM
  Placebo: Placebo comparator
- ETI-204: IM
  ETI-204: monoclonal antibody
- Total: Total of all reporting groups
Arm/Group | Placebo | ETI-204 | Total
Number analyzed (Participants) | 9 | 27 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (11.53) | 47.4 (14.31) | 47.0 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 3 | 16 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 7 | 21 | 28
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 13 | 17
  White | 5 | 12 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Body weight [Mean (Standard Deviation); unit: kg] | 67.71 (13.406) | 76.33 (12.351) | 74.2 (12.989)
Height [Mean (Standard Deviation); unit: cm] | 164.18 (8.859) | 171.01 (8.062) | 169.3 (8.672)
BMI [Mean (Standard Deviation); unit: kg/m2] | 24.92 (2.983) | 26.04 (3.454) | 25.76 (3.337)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Adverse Events
Description: Safety was assessed for all subjects in the Safety Population by collecting and monitoring vital signs, clinical laboratory tests, ECGs, physical examinations, injection site assessments, skin assessments for presence/absence of rash, and adverse events (AEs).
Time Frame: Up to 71 (+/- 4) days or for 30 additional days after the final study visit for subjects with ongoing adverse events at the final scheduled study visit, for each group.
Population: All subjects who received either ETI-204 or placebo were included in the Safety Population. Placebo subject were included in each cohort (one in Cohort 1 and two each in Cohorts 2, 3 ,4 and 5). Safety data are summarized separately for subjects who received ETI-204 in each dose group and for the pooled placebo group.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: ETI-204 placebo IM
- Cohort 1: 4 mg/kg ETI-204 IM
- Cohort 2: 8 mg/kg ETI-204 IM
- Cohort 3: 16 mg/kg ETI-204 IM
- Cohort 4: 20 mg/kg ETI-204 IM
- Cohort 5: 24 mg/kg ETI-203 IM
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 9 | 3 | 6 | 6 | 6 | 6
Participants | 5 | 3 | 1 | 1 | 2 | 2

2. Secondary Outcome: Maximum Observed Plasma Concentration of ETI-204 (Cmax)
Description: Blood samples were obtained and serum concentrations were determined for free ETI-204 using a validated enzyme-linked immunosorbent assay method with an assay range of 100 ng/mL to 5000 ng/mL.
Time Frame: Pre-dose and 1.5, 4, 8, 24, 36, 48, 72 hours after the IM injection of ETI-204 on Day1, and on Days (7), 10, 15, 29, 43, and 71. A Day 7 sample was not included in the profile until the dose had escalated to 20 mg/kg.
Population: The Pharmacokinetic (PK) Population consisted of all subjects who received ETI-204 IM and had at least one valid PK parameter. One subject in Cohort 2 was excluded from the PK Population because the dosing record was missing.
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Cohort 5: 24 mg/kg ETI-204 IM
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 3 | 5 | 6 | 6 | 6
µg/mL | 24.9 (4.70) | 54.8 (6.45) | 105 (22.5) | 118 (28.2) | 154 (32.4)

3. Secondary Outcome: Time to Maximum Observed Plasma Concentration of ETI-204 (Tmax)
Description: as for outcome 2
Time Frame: Pre-dose and 1.5, 4, 8, 24, 36, 48, 72 hours after the IM injection of ETI-204 on Day 1, and on Days (7), 10, 15, 29, 43, and 71. A Day 7 sample was not included in the profile until the dose had escalated to 20 mg/kg.
Population: The PK Population consisted of all subjects who received ETI-204 IM and had at least one valid PK parameter. One subject in Cohort 2 was excluded from the PK Population because the dosing record was missing.
Measure: Median (Full Range); unit: days
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 3 | 5 | 6 | 6 | 6
days | 9.00 [3.00 to 9.00] | 9.00 [3.00 to 9.00] | 6.00 [6.00 to 14.00] | 6.00 [6.00 to 14.00] | 6.00 [3.00 to 9.00]

4. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to Time of Last Quantifiable Concentration (AUC0-last)
Description: as for outcome 2
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µg.day/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 3 | 5 | 6 | 6 | 6
µg.day/mL | 774 (92.3) | 1540 (328) | 2890 (578) | 3660 (945) | 3740 (570)

5. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUC0-inf)
Description: as for outcome 2
Time Frame: as for outcome 3
Population: The PK Population consisted of all subjects who received ETI-204 IM and had at least one valid PK parameter. 1 subject in Cohort 2 was excluded because the dosing record was missing. For 4 subjects (1 in Cohort 2, 1 in Cohort 4. and 2 in Cohort 5) the extrapolated portion of AUC0-inf was >20%; therefore, AUC0-inf was not recorded.
Measure: Mean (Standard Deviation); unit: µg.day/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 3 | 4 | 6 | 5 | 4
µg.day/mL | 819 (85.9) | 1580 (441) | 3200 (755) | 4220 (1360) | 3960 (823)

6. Secondary Outcome: Half-life (t1/2)
Description: as for outcome 2
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 3 | 5 | 6 | 6 | 6
days | 16.0 (1.60) | 20.2 (8.47) | 19.6 (4.10) | 23.3 (6.17) | 20.0 (7.20)

7. Secondary Outcome: Apparent Clearance (CL/F)
Description: as for outcome 2
Time Frame: as for outcome 3
Population: The PK Population consisted of all subjects who received ETI-204 IM and had at least one valid PK parameter.1 subject in Cohort 2 was excluded because the dosing record was missing. For 4 subjects (1 in Cohort 2, 1 in Cohort 4, and 2 in Cohort 5) the extrapolated portion of AUC0-inf was >20%; therefore, AUC0-inf-based parameters were not recorded.
Measure: Mean (Standard Deviation); unit: Liters/day
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 3 | 4 | 6 | 5 | 4
Liters/day | 0.410 (0.0545) | 0.415 (0.117) | 0.445 (0.113) | 0.382 (0.0736) | 0.478 (0.202)

8. Secondary Outcome: Number of Participants With Anti-ETI-204 Antibodies
Description: Blood samples were collected and serum samples were assayed at an initial dilution of 1:10. Samples that were positive at the 1:10 dilution were serially diluted 1:2 and assayed until a negative result was attained. The titer of the most dilute sample yielding a positive result was recorded as the titer for that time point. Immunogenicity was measured by the number of participants in each study arm with anti-ETI-204 antibody values at Days 8, 43 or 71 ≥ 4-times higher than at baseline, or if the titer was negative at baseline, the post-treatment sample(s) required a titer of at least 1:20 for it to be considered positive.
Time Frame: Pre-dose and on Days 10, 43, and 71 after the IM injection of ETI-204 or placebo on Day 1.
Population: All subjects in the Safety Population who received either ETI-204 IM or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 9 | 3 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 71 (+/- 4) days or for 30 additional days after the final scheduled study visit for subjects with ongoing adverse events at that visit, for each group.
Description: Monitoring of Vital signs, clinical laboratory values, ECGs, physical examinations, and adverse events at each scheduled study visit. Skin assessment for presence or absence of rash was performed predose and 1, 2, 4, 12, 24, 48, and 72 hours after the IM injection on Day 1. A Visual Analog Scale for self-evaluation of pain was administered within 0-5 minutes after the IM injection on Day 1 and 2, 4, 8, 24, 48 and 72 hours after the injection.
Groups:
- Cohort 2: 8 mg ETI-204 IM
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/9 | 3/3 | 1/6 | 1/6 | 2/6 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | Cohort 1 (N=3) | Cohort 2 (N=6) | Cohort 3 (N=6) | Cohort 4 (N=6) | Cohort 5 (N=6)
Dizziness (Nervous system disorders) | 0 | 0 (0) | 0 (0) | 0 (0) | 1 | 1
Injection site pain (General disorders) | 2 | 1 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Lip Blister (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Menstruation Irregular (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Procedural Dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tooth Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data generated in this clinical study are the exclusive property of the Sponsor. Written approval from the Sponsor is required prior to disclosing any information related to this clinical study.